CLINICAL TRIAL: NCT04536493
Title: Comparison of 2 Application Techniques for LET (Lidocaine 4%; Epinephrine 0.1%; Tetracaine 0.5%) Gel Used Prior to Simple Laceration Repair
Brief Title: Comparison of 2 Application Techniques for LET Gel Used Prior to Simple Laceration Repair
Acronym: LET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Theodore Heyming, Physician; Emergency Department Medical Director, Children's Hospital of Orange County
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190224
Record Dates: First submitted 2019-06-20; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: LET; Laceration of Skin
MeSH Terms: interventions — Linear Energy Transfer; Tetracaine; Gels

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing two different applications of LET gel in pediatric patients with minor lacerations.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Topical anesthetic applied by RN not involved in procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 application (Active Comparator): Patients receive single dose LET
  Interventions: Drug: LET (lidocaine 4%; epinephrine 0.1%; tetracaine 0.5%) gel (1 application)
- 3 applications (Active Comparator): Patients receive 3 doses of LET
  Interventions: Drug: LET (lidocaine 4%; epinephrine 0.1%; tetracaine 0.5%) gel (3 applications)

INTERVENTIONS:
Drug: LET (lidocaine 4%; epinephrine 0.1%; tetracaine 0.5%) gel (1 application) — 1 application of LET topical anesthetic gel
  Other Names: LET gel
  Arms: 1 application
Drug: LET (lidocaine 4%; epinephrine 0.1%; tetracaine 0.5%) gel (3 applications) — 3 applications of LET topical anesthetic gel
  Other Names: LET gel
  Arms: 3 applications

SUMMARY:
To compare pain scores during laceration repair with first suture placement using standardized visual analog scale (VAS) between 2 different topical local anesthetic application techniques for using LET gel. Specifically, the investigators are studying if applying LET gel 3 times, spaced 10 minutes apart (triple LET) provides superior anesthesia to one 30 minute application (single LET). Single LET is the current standard method of application.

DETAILED DESCRIPTION:
To compare pain scores during laceration repair with first suture placement using standardized visual analog scale (VAS) between 2 different topical local anesthetic application techniques for using LET gel. Specifically, the investigators are studying if applying LET gel 3 times, spaced 10 minutes apart (triple LET) provides superior anesthesia to one 30 minute application (single LET).

Secondary endpoints:

1. To compare provider satisfaction scores using a Likert scale between the triple LET and single LET application techniques.
2. To compare parental satisfaction scores using a Likert scale between the triple LET and single LET application techniques.
3. To compare the need for additional local anesthetic infiltration between the triple LET and single LET application techniques.

Once patients are identified and consent is obtained, they will be randomized to one of two groups. One group will have LET gel applied to the laceration one time for a duration of 30 minutes. The other group will have LET gel applied 3 times, at 10 minute intervals. Between applications, the excess gel on the surface of the skin will be gently wiped off, and a new strip of LET gel will be applied. The laceration repair will proceed in a normal sterile fashion, using standard irrigation and debridement techniques. Laceration repair will occur within the 15 minutes following the 30 minute period of LET application to the wound. The patient will be asked to rate his/her pain immediately after the first suture is placed or attempted using the visual analogue scale (VAS, range 0-10). The decision to use any additional anesthetic infiltration will be left to the performing provider. There will be 2 nurses involved in the study. One nurse will be the patient's primary nurse and will be administering the LET gel (so will not be blinded, but will not be involved in data collection). The other nurse will be obtaining the VAS immediately (Appendix 3) after the first suture is placed, using a pre-prepared script (Appendix 3) and standardized technique. The nurse or research assistant will also be blinded as to the method of LET gel application. The provider performing the laceration repair will be blinded. The research assistant will not be blinded and will coordinate all involved providers and nurses, will ensure correct timing in LET gel administration, and laceration repair timing.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with simple (< 3 cm) lacerations who are > 7 years old and < 18 years old, for whom the physician plans to close the laceration using simple superficial interrupted sutures.

Exclusion Criteria:

* • Lacerations involving the hands, feet, genitals, tongue, mucus membranes, nose, ears, or occurring over joints.

  * Patients who are developmentally delayed or have a disability preventing them from giving a reliable pain score.
  * Patients whose primary language is other than English or Spanish.
  * Patients for whom procedural sedation is required.
  * Patients receiving intranasal or oral midazolam or inhaled nitrous oxide.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
To compare pain scores | The VAS to rate pain will be collected during laceration repair, immediately after the first suture placement or attempt. The VAS score is estimated to take up to 1 minute to collect. The VAS scale will be collected for each enrolled subject.
  Visual Analog Scale (VAS) asks subjects to rate pain marking an X on a line between two ends: "No pain" (on the left) and "Pain as bad as it could possibly be" (on the right). The distance will be measured from "No pain" to the X placed by the subject. A higher measurement indicates more pain.

SECONDARY OUTCOMES:
To compare provider satisfaction scores | The provider satisfaction Likert scale will be collected immediately after the procedure.
  Likert scale will be used in 3 questions asking providers to rate their satisfaction, preference for Single LET application, and preference for Triple LET application. For the satisfaction question, the likert scale offers options from Dissatisfied to Extremely Satisfied, as well as Not Applicable. The preference for Single LET is a likert scale with options ranging from Strongly Disagree to Strongly Agree, as well as a Not Applicable. The preference for Triple LET is a likert scale with options ranging from Strongly Disagree to Strongly Agree, as well as a Not Applicable. It will take approximately 3 minutes to administer. This measure will be completed once for each enrollment prior to discharge from the Emergency Department.
To compare parental satisfaction scores | The parental satisfaction Likert scale will be collected immediately after the procedure.
  Parent satisfaction will be measured using a single question as a Likert scale with options from Dissatisfied to Extremely Satisfied, as well as Not Applicable. It will take approximately 1-2 minutes to administer. This measure will be completed once for each enrollment prior to discharge from the Emergency Department.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Siembieda, Principal Investigator — CHOC Childrens
Locations (1):
- CHOC Children's, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harman S, Zemek R, Duncan MJ, Ying Y, Petrcich W. Efficacy of pain control with topical lidocaine-epinephrine-tetracaine during laceration repair with tissue adhesive in children: a randomized controlled trial. CMAJ. 2013 Sep 17;185(13):E629-34. doi: 10.1503/cmaj.130269. Epub 2013 Jul 29. PMID 23897942
- [Background] Priestley S, Kelly AM, Chow L, Powell C, Williams A. Application of topical local anesthetic at triage reduces treatment time for children with lacerations: a randomized controlled trial. Ann Emerg Med. 2003 Jul;42(1):34-40. doi: 10.1067/mem.2003.207. PMID 12827121